CLINICAL TRIAL: NCT06123754
Title: A Randomized, Controlled, Double-blind, Multicenter Phase III Clinical Study of Envafolimab Plus Platinum-based Doublet Chemotherapy Versus Placebo Plus Platinum-based Doublet Chemotherapy in Patients With Non-small Cell Lung Cancer
Brief Title: Phase III Study of Envafolimab Versus Placebo Plus Chemotherapy in Resectable Stage III NSCLC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: 3D Medicines (Sichuan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: 3D Medicines (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KN035-CN-017
Record Dates: First submitted 2023-10-25; First posted 2023-11-09 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Envafolimab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: This study is a randomized, controlled, double-blind, multicenter phase Ⅲ study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Envalfolimab plus platinum-based doublet chemotherapy (Experimental): Envalfolimab plus platinum-based doublet chemotherapy for a total of 3-4 cycles of neoadjuvant therapy (determined by the investigator), Envafolimab will be administered after surgery at 600 mg every 3 weeks(Q3W) for 16 cycles at most.
  Interventions: Drug: Envalfolimab subcutaneously injected+Platinum-based doublet chemotherapy intravenous injection
- Placebo plus platinum-based doublet chemotherapy (Active Comparator): Placebo plus platinum-based doublet chemotherapy for a total of 3-4 cycles of neoadjuvant therapy (determined by the investigator), placebo will be administered after surgery every 3 weeks(Q3W) for 16 cycles at most.
  Interventions: Drug: placebo subcutaneously injected +Platinum-based doublet chemotherapy intravenous injection

INTERVENTIONS:
Drug: Envalfolimab subcutaneously injected+Platinum-based doublet chemotherapy intravenous injection — The subjects receive Envafolimab/placebo treatment with a dosage of 600 mg/3 ml subcutaneously injected every 3 weeks.It will last about 3-4 cycles before surgery and 16 cycles after surgery.
  Other Names: Experimental
  Arms: Envalfolimab plus platinum-based doublet chemotherapy
Drug: placebo subcutaneously injected +Platinum-based doublet chemotherapy intravenous injection — The subjects received platinum-based doublet chemotherapy on day 1 of every cycle. It's 3 weeks per cycle and lasts 3-4 cycles before surgery.
  Other Names: Active Comparator
  Arms: Placebo plus platinum-based doublet chemotherapy

SUMMARY:
This is a randomized, controlled, double-blind, multicenter Phase 3 clinical study to assess the efficacy and safety of envafolimab plus platinum-based doublet chemotherapy versus placebo plus platinum-based doublet chemotherapy as neoadjuvant/adjuvant therapy in subjects with resectable stage IIIA and IIIB (N2) NSCLC. Primary study endpoints are MPR rate assessed by BIPR and EFS assessed by BIRC.

DETAILED DESCRIPTION:
A total of approximately 390 participants are planned to be enrolled in this study. After being screened and qualified, the subjects will be randomly assigned to receive Envalfolimab or placebo plus platinum-based doublet chemotherapy in 1:1 ratio for a total of 3-4 cycles of neoadjuvant therapy (determined by the investigator), the feasibility of surgery is evaluated by the investigator within 4-6 weeks after the end of neoadjuvant therapy and surgery will be performed. Envafolimab (experimental group) or placebo (control group) will be administered after surgery. After completion of treatment, subjects will enter a follow-up phase, including safety follow-up, tumor disease follow-up, and survival follow-up.All randomized subjects in this study are required to receive tumor imaging evaluation as scheduled and get continuous safety assessment during the srceening and treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate and sign the informed consent form.
2. Age ≥ 18 years old, regardless of gender.
3. Histological and/or cytological diagnosis of resectable stage IIIA-IIIB (N2) NSCLC.
4. Measurable lesions based on the response evaluation criteria in solid tumors version 1.1（RECIST 1.1）.
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
6. Subjects should provide tumor tissue for detection of PD-L1 expression level.
7. Sufficient organ and bone marrow function.
8. Expected survival ≥6 months.
9. The surgeon assessed that total lung function is able to withstand the proposed pneumonectomy procedure.

Exclusion Criteria:

1. Tumor histologically or cytologically confirmed or combined with neuroendocrine carcinoma components, or sarcomatous/sarcomatoid lesions, or adenosquamous carcinoma, or special pathological types.
2. Previous treatment with another drug that targets T cell receptors (e.g. CTLA-4, OX-40, etc.);
3. Participants with known EGFR mutation or ALK translocation, and non-squamous cell carcinoma subjects need to identify EGFR and ALK mutation status;
4. Upper lung sulcus tumor or locally advanced unresectable or metastatic disease.
5. Previous anti-tumor therapy for the disease.
6. Subjects with known or suspected interstitial pneumonia.Radiation pneumonia or other moderate to severe lung disease that may interfere with the detection or management of drug-related pulmonary toxicity and seriously affect respiratory function.
7. Any serious active infection.
8. With uncontrolled or significant cardiovascular and cerebrovascular disease.
9. Active autoimmune disease requiring systemic treatment.
10. Immunosuppressant or systemic hormone therapy (dose >10 mg/ day prednisone or other therapeutic hormone) for immunosuppression within 14 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
MPR by BIPR | Up to 5 years
  MPR rate is defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes following completion of neoadjuvant therapy (evaluated by BIPR)
EFS by BIRC | Up to 5 years
  EFS is defined as the time from randomization until the occurrence of events leading to inoperable disease progression, post-operative disease progression (BIRC assessment based on RECIST 1.1) or recurrence/metastasis, or death from any cause.

SECONDARY OUTCOMES:
pCR | Up to 5 years
  pCR rate is defined as the percentage of participants having an absence of residual invasive cancer in resected lung specimens and lymph nodes following completion of neoadjuvant therapy, assessed by BIPR;
DFS | Up to 5 years
  DFS is defined as the time from post-surgery to radiographic disease progression, local or distant recurrence, or death from any cause, assessed by BIRC;
OS | Up to 5 years
  OS is defined as the time from randomization until death from any cause.;
EFS | Up to 5 years
  EFS is defined as the time from randomization until the occurrence of events leading to inoperable disease progression, post-operative disease progression or recurrence/metastasis, or death from any cause., assessed by investigator;
Explore the quality of life for subjects by EORTC QLQ-C30 | Up to 5 years
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
  Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Explore the quality of life for subjects by EORTC QLQ-LC13 | Up to 5 years
  All of the scales and single-item measures range in score from 0 to 100. A high score for the scales and single items represents a high level of symptomatology or problems.
PD-L1, ctDNA | Up to 5 years
  To explore the correlation between clinical efficacy and tumor tissue sample biomarkers (such as PD-L1 level, etc.) and blood sample biomarkers (such as ctDNA level, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Changli Wang, Principal Investigator — Tianjin Cancer Hospital
Locations (1):
- Tianjin cancer hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided